CLINICAL TRIAL: NCT06717984
Title: A Study on Artificial Intelligence Algorithms for Breast Cancer Classification From Histopathology Images
Brief Title: AI Model for Classifying Breast Cancer From Histopathology Images
Status: Recruiting | Type: Observational
Sponsor: Taufiq Hasan, PhD (Other)
Collaborators: National Institute of Cancer Research & Hospital, Bangladesh (Unknown)
Responsible Party: Sponsor-Investigator, Taufiq Hasan, PhD, Professor, Bangladesh University of Engineering and Technology
Organization: Bangladesh University of Engineering and Technology (Other)
Other Study IDs: NICRH/IRB/2024/134
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Histopathology; Deep Learning
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women who undergo biopsy for suspected abnormal cell growth in the breast: The cohort includes women who have undergone a biopsy due to suspected abnormal cell growth in the breast. This cohort captures a wide range of potential diagnoses, including benign conditions, noninvasive (in situ) breast cancers, and invasive breast cancers. All participants have histopathological samples collected for analysis, which serve as the basis for determining the presence and type of abnormal cell growth. The cohort will be studied using deep learning techniques to classify the biopsy samples into specific categories (normal, benign, in situ, or invasive), with the goal of improving diagnostic accuracy and efficiency in detecting breast cancer.
  By focusing on women undergoing biopsy, this study aims to address the diagnostic challenges faced in distinguishing between various breast tissue abnormalities, contributing to earlier detection and better clinical outcomes.
  Interventions: Diagnostic Test: Biopsy, Mastectomy, Histopathology

INTERVENTIONS:
Diagnostic Test: Biopsy, Mastectomy, Histopathology — Biopsy:
  This intervention involves the collection of breast tissue samples through a biopsy procedure. These samples are obtained from women undergoing investigation for unusual cell growth and are analyzed to detect potential abnormalities, including benign, in situ, or invasive cancerous changes.
  Mastectomy:
  This intervention refers to the surgical removal of breast tissue, typically performed to treat or prevent the spread of breast cancer. It may involve the removal of part or all of the breast and is considered in cases of invasive breast cancer or high-risk noninvasive breast cancer.
  Histopathology:
  This intervention focuses on the microscopic examination of breast tissue samples collected through biopsy or mastectomy. Histopathological analysis is conducted to assess cellular abnormalities, determine the presence of cancer, and classify the tissue as benign, in situ, or invasive, providing the basis for diagnosis and treatment decisions.

SUMMARY:
Breast cancer, a prevalent and potentially fatal disease, underscores the need for early and accurate detection to improve patient outcomes. Traditional histopathological examination, the current gold standard for diagnosis, faces limitations like subjectivity and low efficiency. In response, this research seeks to revolutionize breast cancer diagnostics by using deep learning techniques to classify invasive and noninvasive breast cancer types from histopathological images. Non-invasive cancers, like DCIS and LCIS, are confined to milk ducts or lobules, while invasive cancers spread to surrounding tissue and make up 70% of cases, often leading to poorer outcomes.

The proposed AI model aims to enhance diagnostic accuracy and efficiency, surpassing manual methods, and providing a scalable solution for diverse healthcare settings. By automating image analysis, the model seeks to democratize cancer screening, making it accessible in underserved populations and adaptable to different resources and equipment. Ultimately, this research aims to advance breast cancer detection, improve patient care, and contribute to better treatment outcomes globally.

DETAILED DESCRIPTION:
Breast cancer, a widespread and potentially fatal illness, emphasizes the urgent requirement for early and precise detection to enhance patient outcomes. The current diagnostic framework, characterized by manual histopathological examination, exhibits inherent drawbacks such as subjectivity and limited throughput. In response, our research aims to transform breast cancer diagnostics by leveraging advanced computational techniques, particularly deep learning. Breast cancer can be classified into two main subtypes: invasive and noninvasive.

Noninvasive breast cancer, often termed in situ breast cancer, is characterized by abnormal cells confined within the milk ducts (ductal carcinoma in situ or DCIS) or lobules (lobular carcinoma in situ or LCIS) without invading surrounding tissues. This type is considered an early stage and typically not life-threatening on its own. Invasive breast cancers are those that spread from the original site (either the milk ducts or the lobules) into the surrounding breast tissue. These constitute approximately 70% of all breast cancer cases and generally have a poorer prognosis compared to the in-situ subtypes.

Medical imaging of breasts can be acquired through various techniques, such as MRI scans, mammography, ultrasound, thermography, computed tomography scans, and histopathology. Among these approaches, the histopathology test serves as the gold standard for the clinical diagnosis of cancer.

The proposed AI model aims to streamline and enhance the analysis of histopathological images for the classification of invasive and noninvasive breast cancer, surpassing conventional methods and providing a reliable means of identifying cancerous regions. This promises to significantly improve the accuracy and efficiency of breast cancer diagnostics, meeting the urgent need for dependable and scalable solutions. By automating the complex process of breast cancer histopathological image analysis, our goal is to democratize screening, making it more accessible and reaching underserved populations. Moreover, our model goes beyond technological innovation; it addresses broader issues of accessibility and scalability, particularly in low-income settings. The research's focus on domain adaptation is crucial, ensuring the model's accuracy and reliability across various health facilities. This involves accommodating differences in resources, equipment, and demographic factors, making it a versatile and adaptable solution for diverse contexts.

In summary, our research not only aims to advance the technological frontier in breast cancer diagnostics but also seeks to drive a transformative change in accessibility, efficiency, and reliability. By developing an AI model that tackles the specific challenges of traditional methods, we aim to make a meaningful impact on breast cancer screening, ultimately leading to early detection, tailored treatment, and improved outcomes for patients worldwide.

ELIGIBILITY:
* Inclusion criteria:

  * Female patients of any age can be selected as subjects.
  * Individuals willing to participate in breast cancer screening.
  * Availability for biopsy examination.
  * Women with no current or prior diagnosis of breast cancer.
  * Availability of relevant medical records for confirmation and comparison purposes.
* Exclusion criteria:

  * Pregnant women are excluded due to potential impacts on screening results and the necessity for special considerations during pregnancy.
  * Individuals with severe medical conditions or circumstances that may render histopathologic examination inappropriate or unsafe are excluded.
  * Patients with conditions that could interfere with the accuracy of screening results are excluded.
  * Follow-up screenings are not included in this study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This study is open to female participants only. The focus is on women who are undergoing breast biopsies or mastectomies due to suspected abnormal cell growth, as breast cancer predominantly affects women.
Study Population: The study population includes women who are undergoing breast biopsies or mastectomies due to suspected abnormal cell growth. Participants are drawn from hospitals and clinics where breast cancer screening and diagnostic procedures are conducted. This population includes individuals with a range of breast conditions, from benign abnormalities to noninvasive (in situ) and invasive breast cancers, representing various stages of breast disease for classification and diagnostic purposes.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-02-11 (Estimated); Study Completion 2025-02-11 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Deep Learning Model in Classifying Breast Tissue as Normal Benign, In Situ, or Invasive. | Measured at the time of histopathological image analysis (within 1 week of biopsy or mastectomy).
  The primary outcome of this study is the diagnostic accuracy of the deep learning model in classifying histopathological images from breast biopsies into three categories: benign, in situ (noninvasive), and invasive breast cancer. Accuracy will be measured by comparing the model's predictions to the ground truth diagnoses determined by expert pathologists.

CONTACTS AND LOCATIONS:
Overall Officials: Taufiq Hasan, PhD, Principal Investigator — Department of Biomedical Engineering, Bangladesh University of Engineering and Technology (BUET), Dhaka - 1205.; Farida Arjuman, FCPS, MCPS, Principal Investigator — Department of Histopathology, National Institute of Cancer Research and Hospital (NICRH)
Locations (1):
- National Institute of Cancer Research & Hospital (NICRH), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT06717984/Prot_ICF_000.pdf